CLINICAL TRIAL: NCT03823274
Title: Multi-center, Prospective, Cohort Study to Evaluate the Relationship of Stroke Recurrence and Anti-platelet Resistance in Ischemic Stroke Patients
Status: Completed | Type: Observational
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: YMC037
Record Dates: First submitted 2019-01-24; First posted 2019-01-30 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Aspirin, Clopidogrel — to evaluate the relationship of stroke recurrence and anti-platelet resistance in ischemic stroke patients receiving aspirin and clopidogrel

SUMMARY:
This cohort study will evaluate the relatiobship of stroke recurrence and anti-platelet resistance in ischemic stroke patients

ELIGIBILITY:
Inclusion Criteria:

1. Men and women over 60 years old at the time of written consent
2. Those admitted to the hospital within 72 hours after acute cerebral infarction and treated with Aspirin 100 mg and Clopidogrel 75 mg
3. Written informed consent voluntarily signed

Exclusion Criteria:

1. Those with evidence other brain lesions such as brain tumors
2. Those who need oral anticoagulants other than vitamin K antagonists or anticoagulant therapy of warfarin
3. Contraindicate to Aspirin or Clopidogrel or allergic to the drug
4. Subjects who are at risk of active pathological bleeding such as digestive ulcer and intracranial hemorrhage
5. Cancer disease that can shorten life expectancy
6. Patient's condition that may interfere with participation in study such as mental illness, mental retardation, dementia, drug abuse, and alcoholism
7. Subjects other than the above unsuitable for this clinical study identified by Investigator

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patient
Sampling Method: Non-Probability Sample
Enrollment: 1011 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-01-03 (Actual)

PRIMARY OUTCOMES:
evaluate the relationship of stroke recurrence and anti-platelet resitance | 12weeks
  To evaluate the relationship of stroke recurrence and anti-platelet resitance in ischemic stroke patients receiving aspirin 10mmg and clopidogrel 75mg for 12weeks

CONTACTS AND LOCATIONS:
Overall Officials: jei Kim, Principal Investigator — Chungnam National Universtity Hospital
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea

REFERENCES:
- [Derived] Kim J, Shin BS, Kim DH, Shin DI, Ahn SH, Kim JG, Ryu SH, Moon HR, Kang HG, Jeong H, Yum KS, Chae HY, Kim DH, Kang K, Kim J. Molecular genomic and epigenomic characteristics related to aspirin and clopidogrel resistance. BMC Med Genomics. 2024 Jun 20;17(1):166. doi: 10.1186/s12920-024-01936-1. PMID 38902747